CLINICAL TRIAL: NCT00256919
Title: A Randomised, Placebo-controlled, Parallel Group Single Dose Study of GW856553 in Patients With Active RA to Investigate the C-Reactive Protein (CRP) Dose Response Relationship
Brief Title: Single Dose Study Of GW856553 On A Protein That Is An Indicator For Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA3103730
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: GW856553; biomarkers; CRP; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW856553

SUMMARY:
This study is designed to compare a range of doses of GW856553 versus placebo on the biomarkers associated with rheumatoid arthritis

ELIGIBILITY:
Inclusion criteria:

* Must have a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology.
* Must have 3 or more swollen or 3 or more tender/painful joints at screening.
* Must be on stable weekly methotrexate (2.5mg-25mg) for at least eight weeks prior to screening.

Exclusion criteria:

* Must not be morbidly obese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP) levels 72 hours post-dose. | 72 hours post-dose.

SECONDARY OUTCOMES:
C-reactive protein (CRP) levels 24 and 48 hours post-dose | 24 and 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Germany (4):
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
- Spain (3):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- Sweden (2):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Uppsala
- Ukraine (5):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv

REFERENCES:
- [Derived] Yang S, Lukey P, Beerahee M, Hoke F. Population pharmacokinetics of losmapimod in healthy subjects and patients with rheumatoid arthritis and chronic obstructive pulmonary diseases. Clin Pharmacokinet. 2013 Mar;52(3):187-98. doi: 10.1007/s40262-012-0025-6. PMID 23254770